CLINICAL TRIAL: NCT02238483
Title: A 12-week Phase IIa, Double-blind, Placebo-controlled, Randomized Study to Investigate the Efficacy and Safety of AZD7624 in COPD Patients With a History of Frequent Acute Exacerbations While on Maintenance Therapy
Brief Title: A Phase IIa Study to Investigate the Efficacy and Safety of AZD7624 in Chronic Obstructive Pulmonary Disease (COPD) Patients While on Maintenance Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2550C00005; 2014-001053-16 (EudraCT Number)
Record Dates: First submitted 2014-09-01; First posted 2014-09-12 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD patients; Exacerbations; ICS; LABA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD7624

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD7624 (Experimental): Active treatment
  Interventions: Drug: AZD7624 1.0 mg
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7624 1.0 mg — Inhaled AZD7624 solution, 11 mg/mL
  Arms: AZD7624
Drug: Placebo — Inhaled placebo solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether AZD7624 can reduce acute Chronic Obstructive Pulmonary Disease (COPD) exacerbations in patients on COPD maintenance therapy with a history of frequent acute exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedures.
* Male and females aged 40-85 years. Females must have a negative pregnancy test at Visit 1, must not be lactating and must be of non-childbearing potential. Males must be surgically sterile or agree to use an acceptable method of contraception for the duration of the study and for 3 months after the last dose of investigational product to prevent pregnancy in a partner.
* A weight of ≥50 kg.
* Diagnosis of COPD for more than 1 year at Visit 1, according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2014 guidelines.
* COPD maintenance treatment with at least ICS/LABA for at least 2 months prior to enrolment to be continued unchanged during the study.
* A post-bronchodilator FEV1/FVC <0.70 and a post-bronchodilator FEV1 ≤70% of the predicted normal value. Documented history of 2 or more moderate to severe COPD exacerbations within 12 months of randomisation, but not within the last 6 weeks before randomisation.
* Current or ex-smokers with a smoking history of at least 10 pack-years.

Exclusion Criteria:

* Involvement in the planning and conduct of the study.
* Previous randomisation in the present study.
* Participation in another clinical study with any investigational medicinal product within 3 months of randomisation. Previously intake of any p38 inhibitor.
* Participation in, or scheduled for an intensive COPD rehabilitation programme at any time during the study.
* Planned in-patient surgery or hospitalisation during the study.
* Significant disease or disorder other than COPD which, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study. Asthma as a primary or main diagnosis according to the Global Initiative for Asthma (GINA) guidelines (GINA 2013) or other accepted guidelines.
* A clinically relevant abnormal findings in clinical chemistry, haematology and urinalysis.
* Plasma myoglobin and CK above the upper reference range of the analysing laboratory at randomization.
* A clinically relevant abnormal findings in physical examination, pulse or blood pressure.
* A positive result on screening for serum hepatitis B hepatitis C and Human Immunodeficiency Virus (HIV).
* History or family history of muscle diseases. Abnormal vital signs, defined as Systolic Blood Pressure (SBP) above 140 mmHg if <60 years of age and above 150 mmHg if ≥60 years of age; Diastolic Blood Pressure (DBP) above 90 mmHg; Pulse <50 or >100 bpm.
* Prolonged QTcF >450 ms or family history of long QT syndrome or sudden death at young age. PR(PQ) interval of clinical significance, PR(PQ) > 250 ms.
* Intermittent AV block of 2nd and 3rd degree or AV dissociation.
* Patients with a QRS duration >120 ms.
* Patients with persistent, and/or recurrent symptomatic tachyarrhythmias, as well as patients with an implantable cardioverter-defibrillator (ICD) or a permanent pacemaker.
* Patients with recent Cardiovascular (CV) events or unstable CV disease or a myocardial infarction or stroke within 6 months of screening. History of hospitalization within 12 months caused by heart failure or a diagnosis of heart failure higher than New York Heart Association (NYHA) class II.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7624.
* Any exacerbation or respiratory infection within 6 weeks of randomization.
* Plasma donation within one month of Visit 1, or any blood donation/blood loss >500 mL during the 3 months prior to Visit 1.
* History of, or current alcohol or drug abuse.
* Treatment with any GCS (apart from prescribed steroids at run-in) within 6 weeks of Visit 3 regardless of indication.
* Treatment with strong CYP3A inhibitors within 4 weeks prior to randomisation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naimish Patel, MD, PhD, Study Director — AstraZeneca R&D Boston; Barry Make, MD, FCCP, FACVPR, Principal Investigator — National Jewish Health, Denver, United States
Locations (38):
- United States (20):
  - Research Site, Los Angeles, California
  - Research Site, Torrance, California
  - Research Site, Denver, Colorado
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Larchmont, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Erie, Pennsylvania
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Kingwood, Texas
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Quilmes
  - Research Site, San Miguel de Tucumán
- Chile (3):
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Talcahuano
- Netherlands (4):
  - Research Site, Assen
  - Research Site, Heerlen
  - Research Site, Nijmegen
  - Research Site, Zutphen
- Research Site, Lima, Peru
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, eManzimtoti
  - Research Site, Johannesburg
  - Research Site, Mount Edgecombe
  - Research Site, Parktown West

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-centre study conducted at 39 study centres in 6 countries: Argentina (37.7% of the patients); United States (34.4%) Peru (9%) Chile (6.6%) The Netherlands (6.1%) and South Africa (6.1%) A seasonal recruitment strategy was undertaken where patients were recruited in the fall and winter months of the geographic locality.
Pre-assignment Details: 327 patients signed informed consent, of which 213 patients were randomised. The majority of the 114 not randomised were screening failures
Units Other Than Participants: Patient
Groups:
- AZD7624: Active treatment 2 x 0.5mg inhalation qd
- Placebo: Matching placebo comparator
Period: Overall Study
Arm/Group | AZD7624 | Placebo
Started | 108; 108 Patient | 105; 105 Patient
Completed | 93; 93 Patient | 91; 91 Patient
Not Completed | 15; 15 Patient | 14; 14 Patient
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Death | 1 | 0
Not completed — Adverse Event | 7 | 3
Not completed — Withdrawn due to physician decision | 1 | 0
Not completed — Completion status not recorded | 1 | 1
Not completed — Illness in family member | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient was excluded from the Full Analysis Set due to lack of source data and GCP compliance issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7624 | Placebo | Total
Number analyzed (Participants) | 107 | 105 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 54 | 103
  >=65 years | 58 | 51 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (8.73) | 64.2 (8.67) | 64.8 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 67 | 69 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 65 | 131
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 85 | 88 | 173
  Other | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to First Moderate to Severe COPD Exacerbation or Early Drop-out Related to Worsening of COPD Symptoms
Time Frame: Up to Week 12 treatment discontinuation visit (in some patients this visit was delayed beyond the planned Day 84, up to maximum of 118 days)
Population: The Full Analysis Set excluded one patient due to lack of source data and GCP compliance issues. One further patient was not included in the analysis due to missing covariate data.
Measure: Median (Full Range); unit: days
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
days | NA [5 to NA] — Too few events were observed in the treatment group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range. | 118.0 [4 to NA] — Too few events were observed for the estimation of the upper limit of the full range.
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; H0: Hazard Ratio (AZD7624/placebo) equals 1 vs. H1: Hazard Ratio does not equal 1; Test type: Superiority or Other; p = 0.2371, Regression, Cox; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.81 to 2.40] — A hazard ratio greater than 1 indicates a higher rate of incidence in the AZD7624 group

2. Secondary Outcome: Annual Event Rate of Moderate and Severe COPD Exacerbations and Early Drop-outs Related to Worsening of COPD Symptoms (i.e. Composite Endpoint, ExDo)
Description: For the production of summary statistics, the annual event rate per subject is calculated, and standardized per a 52-week period according to the formula described below.
  Annual Event Rate = No. of Events*365.25 / (Follow-up date - Date of randomization + 1).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Events / year
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
Events / year | 2.16 (0.80) | 1.62 (0.63)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.249, regression, negative binomial; Rate Ratio = 1.33, 95% CI 2-sided [0.82 to 2.16], Standard Error of Mean 0.33 — A hazard ratio greater than 1 indicates a higher rate of incidence in the AZD7624 group

3. Secondary Outcome: Time to First Event of Moderate or Severe COPD Exacerbations or Early Drop-out (Including Drop-outs Due to Any Cause)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
days | NA [5 to NA] — Too few events were observed in the treatment group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range. | 118.0 [4 to NA] — Too few events were observed for the estimation of the upper limit of the full range.
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.1261, Regression, Cox; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.89 to 2.50] — A hazard ratio greater than 1 indicates a higher rate of incidence in the AZD7624 group

4. Secondary Outcome: Annual Event Rate of Moderate and Severe COPD Exacerbations and Early Drop-outs (Including Drop-outs Due to Any Cause)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Events / year
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
Events / year | 2.17 (0.80) | 1.55 (0.60)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.157, regression, negative binomial; Rate ratio = 1.40, 95% CI 2-sided [0.88 to 2.21], Standard Error of Mean 0.33

5. Secondary Outcome: Time to First Moderate or Severe Exacerbation
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
days | NA [5 to NA] — Too few events were observed in the treatment group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range. | NA [4 to NA] — Too few events were observed in the placebo group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range.
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.1529, Regression, Cox; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [0.85 to 2.76]

6. Secondary Outcome: Annual Exacerbation Rate of Moderate and Severe Exacerbations
Description: For the production of summary statistics, the annual exacerbation rate per subject is calculated, and standardized per a 52-week period according to the formula described below.
  Annual Exacerbation Rate = No. of Exacerbations*365.25 / (Follow-up date - Date of randomization + 1).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Exacerbations / year
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
Exacerbations / year | 2.12 (0.78) | 1.42 (0.56)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.129, regression, negative binomial; rate ratio = 1.50, 95% CI 2-sided [0.89 to 2.52], Standard Error of Mean 0.40

7. Secondary Outcome: Time to First Moderate or Severe Exacerbation (Where Worsening of COPD Symptoms is Defined as Anthonisens Criteria Fulfilled)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
days | NA [6 to NA] — Too few events were observed in the treatment group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range. | NA [4 to NA] — Too few events were observed in the placebo group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range.
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.8543, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.43 to 2.01] — A hazard ratio greater than 1 indicates a higher rate of incidence in the AZD7624 group

8. Secondary Outcome: Annual Exacerbation Rate of Moderate and Severe Exacerbations (Where Worsening of COPD Symptoms is Defined as Anthonisens Criteria Fulfilled)
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Exacerbations / year
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
Exacerbations / year | 1.23 (0.39) | 1.09 (0.37)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.751, regression, negative binomial; rate ratio = 1.12, 95% CI 2-sided [0.55 to 2.29], Standard Error of Mean 0.41

9. Secondary Outcome: Time to First Symptom Defined Exacerbation (as Defined by the Exacerbation of Chronic Pulmonary Disease Tool [EXACT] Daily Diary)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
days | NA [3 to NA] — Too few events were observed in the treatment group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range. | NA [2 to NA] — Too few events were observed in the placebo group for the estimation of median using Kaplan-Meier methodology. Too few events were observed for the estimation of the upper limit of the full range.
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.5381, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.54 to 1.38] — A hazard ratio greater than 1 indicates a higher rate of incidence in the AZD7624 group

10. Secondary Outcome: Annual Exacerbation Rate of Symptom Defined Exacerbations (as Defined by the EXACT Daily Diary)
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Exacerbations / year
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
Exacerbations / year | 1.96 (0.54) | 2.33 (0.64)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.440, regression, negative binomial; rate ratio = 0.84, 95% CI 2-sided [0.55 to 1.30], Standard Error of Mean 0.19

11. Secondary Outcome: Symptoms of COPD (Using the EXACT for Respiratory Symptoms [E-RS] Total Score, a Subset of Items From the EXACT Diary)
Description: The EXACT for Respiratory Symptoms (E-RS) scale is a derivative instrument comprising a subset of 11 of the EXACT items to evaluate the severity of respiratory symptoms of COPD. Summation of E-RS item responses produces a total score ranging from 0 to 40, with higher scores indicating greater severity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 106 | 105
scores on a scale | -0.21 (0.88) | 0.17 (0.91)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.5474, Mixed Models Analysis; Mean Difference (Net) = -0.37, 95% CI 2-sided [-1.60 to 0.85] — LSMean difference for overall treatment effect. Negative values for a difference show AZD7624 to have a favourable outcome compared to Placebo

12. Secondary Outcome: Health Related Quality of Life (as Assessed by St Georges Respiratory Questionnaire for COPD Patients [SGRQ-C])
Description: The SGRQ-C is a modified version of the St. George's Respiratory Questionnaire, which has been developed to measure the impact of respiratory disease on health status. The SGRQ-C includes 14 questions in 3 domains: symptoms; activity; and impacts. Scores range from 0 to 100 with higher scores indicating benefit. Change in total score from pre study-treatment baseline to Week 12 end of treatment visit are reported.
Time Frame: as for outcome 1
Population: Full Analysis Set excluding one patient due to lack of source data and GCP compliance issues.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 107 | 105
scores on a scale | -4.03 (19.574) | -5.11 (17.809)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.6352, Mixed Models Analysis; Mean Difference (Net) = 0.83, 95% CI 2-sided [-2.62 to 4.29] — LSMean difference for overall treatment effect. Positive values for a difference show AZD7624 to have a favourable outcome compared to Placebo

13. Secondary Outcome: Dyspnea (Transitional Dyspnea Index (TDI) Score)
Description: The Baseline/Transitional Dyspnea Index (BDI/TDI) provides a multidimensional measure of dyspnea in relation to activities of daily living. The BDI provides a measure of dyspnoea at a single state, the baseline, and the TDI evaluates changes in dyspnoea from the baseline state. The instrument consists of three components: functional impairment, magnitude of task, and magnitude of effort. For the BDI, each of these three components are rated in five grades from 0 (severe) to 4 (unimpaired), and are summed to form a baseline total score from 0 to 12. For the TDI, changes in dyspnea are rated for each component by seven grades from -3 (major deterioration) to +3 (major improvement), and are added to form a total TDI score from -9 to +9. Positive scores indicate an improvement, and a change from the BDI or a difference between treatments of 1 point has been estimated to constitute the minimum clinically important difference.
Time Frame: as for outcome 1
Population: The Full Analysis Set excluded one patient due to lack of source data and GCP compliance issues. Only patients with post-baseline TDI scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 102 | 100
score on a scale | 0.41 (0.15) | 0.54 (0.16)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.2694, Mixed Models Analysis; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.34 to 0.10] — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Pulmonary Function Measured as Changes From Baseline (Post-bronchodilator at Visit 3) in Trough Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: as for outcome 1
Population: Full Analysis Set excluding one patient due to lack of source data and GCP compliance issues.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 107 | 105
Litres | -0.003 (0.2555) | -0.028 (0.2317)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.5144, Mixed Models Analysis; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.03 to 0.07] — [estimate comment as in outcome 12, analysis 1]

15. Secondary Outcome: Pulmonary Function Measured as Changes From Baseline (Post-bronchodilator at Visit 3) in Trough Forced Vital Capacity (FVC)
Time Frame: as for outcome 1
Population: Full Analysis Set excluding one patient due to lack of source data and GCP compliance issues.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 107 | 105
Litres | -0.045 (0.4017) | -0.018 (0.3890)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.5416, Mixed Models Analysis; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.10 to 0.05] — [estimate comment as in outcome 12, analysis 1]

16. Secondary Outcome: Pulmonary Function Measured as Changes From Baseline (Post-bronchodilator at Visit 3) in Trough FEV1/FVC Ratio
Time Frame: as for outcome 1
Population: Full Analysis Set excluding one patient due to lack of source data and GCP compliance issues.
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | AZD7624 | Placebo
Number analyzed (Participants) | 107 | 105
L/L | 0.0077 (0.05269) | -0.0072 (0.05255)
Statistical Analysis 1: Comparison: AZD7624 vs Placebo; Test type: Superiority or Other; p = 0.1965, Mixed Models Analysis; Mean Difference (Net) = 0.01, 95% CI 2-sided [0.00 to 0.02] — [estimate comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from informed consent throughout the study until follow-up (Week 14). Adverse events (AEs) were collected from Visit 2 (start of OCS treatment) throughout the study until follow-up (Week 14).
Arm/Group | AZD7624 | Placebo
Serious Adverse Events (participants affected / at risk) | 11/108 | 11/105
Other Adverse Events (participants affected / at risk) | 71/108 | 48/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7624 (N=108) | Placebo (N=105)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7624 (N=108) | Placebo (N=105)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 31 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Dysgeusia (Nervous system disorders) | 5 | 1
Influenza (Infections and infestations) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Bronchitis (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4
Fatigue (General disorders) | 3 | 0
Hypertension (Vascular disorders) | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Asthenia (General disorders) | 2 | 4
Sinusitis (Infections and infestations) | 1 | 3
Oedema peripheral (General disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No